CLINICAL TRIAL: NCT03089151
Title: A Pilot Randomized Controlled Trial of Gardening as an Intervention to Reduce Risk of Cancer and Heart
Brief Title: Denver Garden Environment and Microbiome Study Disease
Acronym: DGEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Jill Litt, Associate Professor, Environmental Studies, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 16-0138, 16-0424
Record Dates: First submitted 2017-02-17; First posted 2017-03-24 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Diet Modification; Physical Activity; Weight Gain; Chronic Disease; Lifestyle, Sedentary; Health Behavior
Keywords: Pilot Randomized Controlled Trial; Community Garden; Health Behavior Change; Physical Activity; Diet; Obesity; Neighborhood; Microbiome; Inflammatory biomarkers
MeSH Terms: conditions — Motor Activity; Weight Gain; Chronic Disease; Sedentary Behavior; Health Behavior; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Garden Intervention Group (Experimental): Participants randomized to the Community Garden Intervention Group will receive the garden intervention. Participants will be assigned a plot for one season and will receive a standard package of services and amenities to support participation in the community garden, including seeds and transplants, tools, new garden classes and access to master community gardeners in Denver.
  Interventions: Behavioral: Community Garden Intervention
- Wait List Control Group (No Intervention): The non-gardening group will remain on the DUG wait lists and will not receive the garden intervention.

INTERVENTIONS:
Behavioral: Community Garden Intervention — The investigators will recruit 30 prospective gardeners who have not been gardening for the past two years and who are listed on Denver Urban Gardens (DUG) wait lists. DUG randomly assigns people on each garden wait list to available plots, using a lottery. This creates a natural randomized experiment. Participants randomized to the garden intervention will receive a standardized garden resource package, which includes the following:
  1. A garden plot in a Denver Urban Garden
  2. Seeds and plant starts
  3. Introductory gardening workshop
  4. Social events including garden-specific events and garden mentoring.
  The non-gardening group will remain on the DUG wait lists and will not receive these resources.
  Duration of the intervention is 1 year.
  Arms: Community Garden Intervention Group

SUMMARY:
An interdisciplinary team with extensive garden study experience conducted a pilot randomized controlled clinical trial to see whether gardening reduced risk factors for diseases like cancer and heart disease. The pilot trial will provide preliminary data on associations between human microbiome, diet, physical activity, and social interactions and the outcomes of weight status and key inflammatory biomarkers.

DETAILED DESCRIPTION:
The pilot study will lead to development of a future, large randomized controlled clinical trial, by fulfilling the following aims:

Pilot Aim 1: Demonstrate feasibility of recruitment and ability to perform study procedures.

Pilot Aim 2: Demonstrate the ability to measure accurately chronic disease risk factors such as diet, physical activity, weight gain, microbiome characteristics and inflammatory biomarkers.

Pilot Aim 3: Provide preliminary results on the efficacy of gardens as a preventive intervention, and estimates for a detailed power analysis for the proposed subsequent larger trial.

Aim 3a: Demonstrate that compared to non-gardeners, gardeners have 1) greater intake of fruits and vegetables; 2) better Healthy Eating Index (HEI); 3) lower Diet Inflammatory Index (DII); 4) reduced sedentary time and increased moderate-to-vigorous physical activity (MVPA); and reduced age-associated weight gain.

Aim 3b: For gardeners and non-gardeners, sample garden soil, gut, skin, and oral microbiome at six time points from April through September to characterize and compare bacterial load, pathogenic taxa, taxonomic diversity, relative dominance, indicator taxa, and metabolomic results.

Aim 3c: Demonstrate that gardening reduces inflammatory biomarkers linked to heart disease and cancer, including CRP, IL1b, IL4, IL6, IL10, and TNFa, and that the effect of gardening is mediated by diet, weight gain, physical activity and characteristics of the microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent in English or Spanish
* Aged 18 or over
* Currently on the wait list for a new garden
* Not have gardened in the past 2 gardening seasons

Exclusion Criteria:

* Is not able to complete the study requirements in Spanish or English
* Aged 17 or younger
* Has gardened in the past 2 gardening seasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Change in fruit and vegetable intake from baseline at 20 weeks | Measurements will occur during weeks 1-2 (3 random recalls) and weeks 18-20 (3 random recalls)
  6 24-hour diet recalls will be collected at random
Change in sedentary time behavior from baseline at 20 weeks | 2 measurements over 6 months, T1 (Week 1) and T6 (Week 20)
  Accelerometers will be adhered to thigh and collect data for 7 days
Change in bacterial load from baseline at 20 weeks | Every 3-4 weeks up to 20 weeks (Week 1, Week 4, Week 7, Week 10, Week 14, Week 18)
  Microbiome data will be collected six time points using 1 gut, 2 skin, and 1 oral samples
Change in moderate-to-vigorous physical activity (MVPA) from baseline at 20 weeks | 2 measurements over 6 months, T1 (Week 1) and T6 (Week 20)
  Accelerometers will be adhered to thigh and collect data for 7 days
Change in weight (kg) from baseline at 20 weeks | 2 measurements over 6 months, T1 (Week 1) and T6 (Week 20)
  Objective measurements of weight will be collected
Change in waist circumference from baseline at 20 weeks | 2 measurements over 6 months, T1 (Week 1) and T6 (Week 20)
  Objective measurement of waist circumference
Change in pathogenic taxa from baseline at 20 weeks | Every 3-4 weeks up to 20 weeks (Week 1, Week 4, Week 7, Week 10, Week 14, Week 18)
  Microbiome data will be derived from 1 gut, 2 skin, and 1 oral samples
Change in taxonomic diversity from baseline at 20 weeks | Every 3-4 weeks up to 20 weeks (Week 1, Week 4, Week 7, Week 10, Week 14, Week 18)
  Microbiome data will be derived from 1 gut, 2 skin, and 1 oral samples
Change in relative dominance from baseline at 20 weeks | Every 3-4 weeks up to 20 weeks (Week 1, Week 4, Week 7, Week 10, Week 14, Week 18)
  Microbiome data will be derived from 1 gut, 2 skin, and 1 oral samples
Change in indicator taxa from baseline at 20 weeks | Every 3-4 weeks up to 20 weeks (Week 1, Week 4, Week 7, Week 10, Week 14, Week 18)
  Microbiome data will be derived from 1 gut, 2 skin, and 1 oral samples
Change in Inflammatory biomarkers from baseline at 20 weeks | 20 weeks
  Samples include hs-CRP, TNF-alpha, IL1b, IL4, IL6, IL10

SECONDARY OUTCOMES:
Change in HbA1C from baseline at 20 weeks | 20 weeks
Change in blood pressure from baseline at 20 weeks | 20 weeks
Change in lipid profile from baseline at 20 weeks | 20 weeks
  Including LDL, HDL, total cholesterol, triglycerides

CONTACTS AND LOCATIONS:
Overall Officials: Jill S Litt, PhD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No